CLINICAL TRIAL: NCT06559722
Title: A 26-Week,Randomised,Open-Label,Multicenter,Active-Controlled,Parallel-Design,Phase III Clinical Trial to Compare the Efficacy and Safety of Insulin Degludec/Liraglutide Injection With XULTOPHY® Once Daily Via Subcutaneous Injection in Chinese Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Efficacy and Safety of Insulin Degludec/Liraglutide Injection in Subjects With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THDB0213L03
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira; Xultophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Degludec/liraglutide injection (Experimental): Subcutaneously (s.c., under the skin) administration once daily in combination with metformin. Dose was individually adjusted.
  Interventions: Drug: Insulin Degludec/liraglutide Injection
- XULTOPHY® (Active Comparator): Subcutaneously (s.c., under the skin)administration once daily in combination with metformin. Dose was individually adjusted.
  Interventions: Drug: XULTOPHY®

INTERVENTIONS:
Drug: Insulin Degludec/liraglutide Injection — Subcutaneously (s.c., under the skin)administration once daily in combination with metformin. Dose was individually adjusted.
  Arms: Insulin Degludec/liraglutide injection
Drug: XULTOPHY® — Subcutaneously (s.c., under the skin)administration once daily in combination with metformin. Dose was individually adjusted.
  Arms: XULTOPHY®

SUMMARY:
This is a randomised, open-label, multicenter, active-controlled, parallel-design, phase III clinical trial. The purpose of this study to compare the efficacy and safety of Insulin Degludec/Liraglutide Injection with XULTOPHY® once daily via subcutaneous injection in Chinese Subjects with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily participate in this clinical trial and signed the informed consent form (ICF);
* Chinese subjects aged 18-75 years (both inclusive) at the time of consent, male or female;
* Type 2 diabetes mellitus (clinically diagnosed for more than 6 months);
* HbA1c7.0-10.0 % (both inclusive) by central laboratory analysis at the time of screening;
* Current treatment for at least 90 calendar days prior to screening with metformin monotherapy or metformin in any combination with 1 additional OADs (including fixed combination): SU, glinides, AGI, SGLT2i or TZD. For ≥ 60 calendar days prior to screening subjects should be on a stable dose of:

  1. Metformin (≥ 1500 mg or at maximum tolerated dose) or
  2. Metformin (≥1500 mg or max tolerated dose) and SU (≥half of the max approved dose according to local label) or
  3. Metformin (≥1500 mg or max tolerated dose) and glinides (≥half of the max approved dose according to local label) or
  4. Metformin (≥1500 mg or max tolerated dose) and AGI (≥half of the max approved dose according to local label) or
  5. Metformin (≥1500 mg or max tolerated dose) and SGLT2i (≥half of the max approved dose or minimum maintenance dose such as empagliflozin 10 mg and canagliflozin 100 mg according to local label) or
  6. Metformin (≥1500 mg or max tolerated dose) and TZD (≥half of the max approved dose according to local label);
* Body mass index (BMI) ≥ 19.0 kg/m2 and ≤ 40 kg/m2;
* Able and willing to adhere to the protocol including performing self-monitoring of plasma glucose profiles, keeping a trial diary and using a pre-filled pen device.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

* Subjects with diabetes of other types than T2DM;
* Known or suspected hypersensitivity to trial product(s) or related components;
* Participated in any clinical trial and Receipt of any treatment of investigational medicinal product (IMP) or medical device within 90 days prior screening;
* Treatment with glucose lowering agent(s) other than stated in the inclusion criteria 5 for cumulatively more than 14 days in a period of 90 days before screening; or treatment with these agent(s) in a period of 30 days before screening and might influence the assessment of efficacy of glycemic control (Judged by the investigator);
* Treatment with systemic corticosteroid for cumulatively more than 14 days in a period of 90 days before screening (including intravenous, muscle and subcutaneous injections, and oral administration, except for local, intraocular, nasal, intraarticular, and inhalation medications); or treatment with these agent(s) in a period of 30 days before screening and might influence the assessment of efficacy (Judged by the investigator);
* Treatment with glucose lowering agent(s) of herbal traditional Chinese medicine or other local herbal medicines for cumulatively more than 14 days in a period of 90 days before screening; or treatment with these agent(s) in a period of 30 days before screening and might influence the assessment of efficacy (Judged by the investigator);
* Treated with stable insulin regimen (except for short-term treatment (e.g., no more than 14 days of continuous treatment)), or treatment with insulin in a period of 30 days before screening and might influence the assessment of efficacy (Judged by the investigator);
* Treatment with GLP-1 receptor agonists or DPP-4 inhibitors within 90 calendar days prior to screening;
* Impaired liver function, defined as aspart aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 times upper limit of the normal or a total bilirubin level (TBIL) ≥ 1.5 times upper limit of the normal;
* Triglycerides >5.6 mmol/L at screening;
* Impaired renal function, defined as creatinine clearance (Ccr) of less than 60 mL/min (calculated from the Cockcroft-Gault formula);
* Have had 1 or more episodes of severe hypoglycemia within the 6 months prior to screening.
* Have had 1 or more episodes of acute diabetic complications (diabetic ketoacidosis, hyperglycemic hyperosmolar state, diabetic lactic acidosis, etc.) within the 6 months prior to screening.
* With concomitant conditions at screening that may affect the evaluation of the study, including cardiovascular and cerebrovascular diseases, respiratory diseases, gastrointestinal diseases, liver diseases, kidney diseases, nervous system diseases, psychiatric diseases, hematological diseases, immune system diseases, endocrine system diseases, pancreatic diseases, and/or malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c after 26 weeks of treatment | Baseline, Week 26
  Calculated based on HbA1c level measured in plasma

SECONDARY OUTCOMES:
Proportion of subjects that achieved HbA1c<7% after 12, 26 weeks of treatment | Week 12, Week 26
  Calculated based on HbA1c level measured in plasma
Proportion of subjects that achieved HbA 1c ≤ 6.5% after 12, 26 weeks of treatment | Week 12, Week 26
  Calculated based on HbA1c level measured in plasma
Changes from baseline in fasting plasma glucose (FPG) after 12, 26 weeks of treatment | Baseline, Week 12, Week 26
  Calculated based on FPG level measured in plasma
Change from baseline in 7-point SMBG values after 12, 26 weeks of treatment | Baseline, Week 12, Week 26
  Calculated based on 7-point SMBG values
Change from baseline in body weight after 12, 26 weeks of treatment | Baseline, Week 12, Week 26
  Calculated based on body weight measurement
Number of treatment emergent adverse events | From Baseline to Week 27
  Count
Number of treatment emergent hypoglycaemic episodes | From Baseline to Week 27
  Count
Number of participants with injection site reactions | From Baseline to Week 27
  Count (spontaneous pain, tenderness, itching, redness, edema, induration/infiltration)
Incidence of anti-drug antibodies (ADA), and neutralising antibodies (if applicable) | Baseline, Week 12, 26, and 27 (if applicable)
  Calculated based on the values of anti-drug antibodies (ADA), and neutralising antibodies (if applicable)
Plasma concentrations of degludec, liraglutide | Baseline, Week 2, 6, 12, 20, 26
  Calculated based on plasma concentrations of degludec, liraglutide